CLINICAL TRIAL: NCT03111979
Title: The Effects of 4 Week β-alanine Supplementation on Knee Extensor Contractile and Force Properties in the Over 60s
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Time restrictions on leading investigator
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Rebecca Louise Jones, Academic Associate, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 343
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Muscle Function
Keywords: beta-alanine; Carnosine; Neuromuscular; Stimulation; Skeletal muscle
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine supplementation (Experimental): Participants will be supplemented with 4.8g·d-1 β-alanine (CarnoSyn™, NAI, USA). The β-alanine dosing regimen will consist of two 800 mg tablets three times per day at 3-4 hour intervals or the same regimen for placebo tablets. The use of multiple small doses throughout the day has been used in numerous studies using β-alanine in solutions or gelatine capsules (Hoffman et al., 2008; Sale et al., 2011; Saunders et al., 2012; Sale et al., 2012; Tobias et al., 2013) in order to circumvent potential symptoms of paraesthesia (see box xii for possible risks and discomforts). Overall increases have been shown to be between 40% and 80% depending upon dose (between 3.2 and 6.4 g·d-1) and duration of administration (between 4 and 10 weeks) (Sale et al., 2012).
  Interventions: Dietary Supplement: beta-alanine
- Placebo (Placebo Comparator): Participants will be supplemented with 4.8 g·d-1 placebo (maltodextrin; NAI, USA). The regimen will consist of two 800 mg tablets three times per day at 3-4 hour intervals the same regimen for beta-alanine tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: beta-alanine
  Arms: Beta-alanine supplementation
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The older population is the fastest growing age group worldwide, but it is also the most susceptible to chronic diseases and disabilities. One of the most common negative consequences of aging is the decline in muscle mass, strength and power. This is most notable in lower limb muscles. These muscles are required for the performance of daily activities including walking, stair climbing and standing up from sitting. Regular exercise is considered one of the most effective measures to slow, and even reverse the progression of muscle weakness. Nevertheless older adults may notice a decline in their capability to undertake regular exercises, this may be due to a decline in their muscle's ability to buffer pH. Carnosine (made by bonding β-alanine and histidine) has been suggested to contribute to the extension of physical performance, counteracting the decline the muscle's ability to buffer pH. Yet this pH buffering process it largely restricted by the amount of β-alanine available in the human body. β-alanine is already known to decline in older individuals due to a reduction in food products (meat, fish and poultry). Yet through either consumption of β-alanine rich food, or through short-term supplementation, β-alanine is raised, increasing carnosine concentrations. Improved β-alanine levels can potentially advance exercise performance, for example significant improvements in time to exhaustion on both a constant (37%) and incremental (12%) treadmill tests have been demonstrated. It is therefore proposed that via β-alanine supplementation, an individual's perception of their frailty, maintenance of health and independent living can be improved in older individuals.

However, these findings are based on participants, both young and older, who are well-rested with no prior exercise or fatigue to the assessed muscles. It remains unclear if β-alanine supplementation will aid in the buffering of pH when the muscle has already been fatigued. Therefore this investigation hopes to examine the effects of 4 week β-alanine supplementation on lower limb contractile and force properties, pre and post muscle specific fatigue.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be defined as 'medically stable' for exercise studies, as proposed by Grieg et al. (1994). This criteria was designed both for safety and to define degrees of freedom from diseases which might alter exercise performance (Greig et al., 1994).

Exclusion Criteria:

* Participants will be excluded if they are vegetarian/vegan or have been using β-alanine or creatine supplements within the past 6 months. They will also be excluded if they have participated in a resistance training programme in the last 6 months. These criteria will apply throughout the whole study, with any participants immediately excluded from the study if any of these medical conditions should arise.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Half relaxation time | 4 weeks
  The time taken to decline to 50% maximum following a evoked twitch contraction

SECONDARY OUTCOMES:
Force frequency relationship | 4 weeks
  Assessed during electrically evoked contractions
Time to peak tension | 4 weeks
  The time taken to reach peak in evoked twitch contractions
Electromechanical delay | 4 weeks
  The time between EMG onset and force onset in twitch contractions
Maximal voluntary force production | 4 weeks
  The maximal force produced during a voluntary isometric contraction
Explosive voluntary force production | 4 weeks
  The quickest rate of force developed during voluntary isometric contractions at greater than 80% of voluntary maximum, with no pre-tension or swinging back of the assessed leg.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sale C, Saunders B, Harris RC. Effect of beta-alanine supplementation on muscle carnosine concentrations and exercise performance. Amino Acids. 2010 Jul;39(2):321-33. doi: 10.1007/s00726-009-0443-4. Epub 2009 Dec 20. PMID 20091069
- [Result] Sale C, Artioli GG, Gualano B, Saunders B, Hobson RM, Harris RC. Carnosine: from exercise performance to health. Amino Acids. 2013 Jun;44(6):1477-91. doi: 10.1007/s00726-013-1476-2. Epub 2013 Mar 12. PMID 23479117
- [Result] Harris RC, Sale C. Beta-alanine supplementation in high-intensity exercise. Med Sport Sci. 2012;59:1-17. doi: 10.1159/000342372. Epub 2012 Oct 15. PMID 23075550
- [Result] Artioli GG, Gualano B, Smith A, Stout J, Lancha AH Jr. Role of beta-alanine supplementation on muscle carnosine and exercise performance. Med Sci Sports Exerc. 2010 Jun;42(6):1162-73. doi: 10.1249/MSS.0b013e3181c74e38. PMID 20479615